CLINICAL TRIAL: NCT03949985
Title: Longitudinal Hemostatic Profile After Stopping Estroprogestative Contraceptives: a Prospective Cohort Study
Brief Title: Longitudinal Hemostatic Profile After Stopping Estroprogestative Contraceptives
Acronym: PILL-OFF
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Marc Blondon, Co-Principal Investigator, University Hospital, Geneva
Other Study IDs: 2018-00448
Record Dates: First submitted 2019-05-08; First posted 2019-05-14 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Venous Thromboembolism; Contraception
MeSH Terms: conditions — Venous Thromboembolism | interventions — Contraceptive Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Estrogenic contraceptive users
  Interventions: Other: Tests of biological hemostatic profile associated with contraceptives
- Non-estrogenic contraceptive users
  Interventions: Other: Tests of biological hemostatic profile associated with contraceptives

INTERVENTIONS:
Other: Tests of biological hemostatic profile associated with contraceptives — Tests of biological hemostatic profile associated with contraceptives will be done before and after having stopped an estrogenic contraceptive (group 1) and during the non-use of an estrogenic contraceptive (group 2)

SUMMARY:
This prospective cohort evaluates the longitudinal profile of hemostatic biomarkers during the first 3 months after having stopped a combined oral contraceptive.

DETAILED DESCRIPTION:
Women using a combined oral contraceptive (COC) and who have decided to stop it or switch it to a non-estrogenic contraceptive are included. At baseline, before the COC is stopped, and at multiple time points during the 3 months of follow-up, blood will be drawn to evaluate the hemostatic profile. Findings are compared with a control group of women without an estrogenic contraceptive, who are also followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* women
* 18-50 years
* current use (for at least 3 months) of an estrogenic contraceptive with the decision to stop it or replace it with a non-estrogenic contraceptive (estrogen group)
* no current use of an estrogenic contraceptive (control group)

Exclusion Criteria:

* personal history of VTE
* known thrombophilia
* recent medical event (hospitalization, surgery, cancer)
* pregnancy, post-partum period, current breastfeeding

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: Women aged 18-50 years who are current users of estrogenic contraceptives and have decided to stop it or replace it with a non-estrogenic contraceptive.
  Women aged 18-50 years who are not current users of estrogenic contraceptives.
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2020-09-14 (Actual); Study Completion 2020-09-14 (Actual)

PRIMARY OUTCOMES:
Change in normalized APC sensitivity ratio | Three months

SECONDARY OUTCOMES:
Change in Endogenous Thrombin Potential (Thrombin Generation Assay) | Three months
Change in concentrations of sex hormone-binding globulin | Three months
Change in fibrinolysis assay | Three months
Change in individual coagulation factors | Three months
  The following coagulation factors will be assessed: fibrinogen, protein C, protein S, antithrombin, factor VIII
Contraception-related satisfaction | Three months
  Satisfaction will be estimated by the use of the Ortho Birth Control Satisfaction Assessment Tool questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Geneva University Hospitals, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hugon-Rodin J, Fontana P, Poncet A, Streuli I, Casini A, Blondon M. Longitudinal profile of estrogen-related thrombotic biomarkers after cessation of combined hormonal contraceptives. Blood. 2024 Jan 4;143(1):70-78. doi: 10.1182/blood.2023021717. PMID 37939264